CLINICAL TRIAL: NCT03479099
Title: Clinical Utility of Combined CTC and ctDNA Assay in the Diagnosis of Primary Lung Cancer
Brief Title: Liquid Biopsy in Lung Cancer
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Sang-Won Um, Associate Professor, Samsung Medical Center
Other Study IDs: 2018-01-081
Record Dates: First submitted 2018-03-12; First posted 2018-03-27 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Lung Cancer (Diagnosis); Circulating Tumor Cell
Keywords: Lung cancer; Circulating Tumor Cell; Cell-Free Tumor DNA; Liquid Biopsy
MeSH Terms: conditions — Lung Neoplasms; Disease; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to assess clinical utility of combined circulating tumor cell (CTC) and circulating tumor DNA (ctDNA) in the diagnosis of primary lung cancer.

DETAILED DESCRIPTION:
The peripheral blood and tumor tissue samples are collected from the participants.CTC and ctDNA are analyzed from the blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histology-proven lung cancer or a clinical suspicion of lung cancer
* Age >=18, < 80 years
* No previous history of cancer treatment within 5 years
* Patients who agree to participate

Exclusion Criteria:

* Patients who have been diagnosed with malignancy within 5 years
* Patients with previous history of lung cancer
* Patients who have uncontrolled coagulopathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects who are referred for the evaluation and management of primary lung cancer in the tertiary care center
Sampling Method: Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-03-11 (Actual)

PRIMARY OUTCOMES:
Diagnostic sensitivity of combined CTC and ctDNA | 1 year
  To compared the sensitivity of combined CTC and ctDNA with those of CTC and ctDNA alone in diagnosis of primary lung cancer

SECONDARY OUTCOMES:
Diagnostic accuracy of combined CTC and ctDNA | 1 year
  To compared the accuracy of combined CTC and ctDNA with those of CTC and ctDNA alone in diagnosis of primary lung cancer
Diagnostic specificity of CTC and ctDNA | 1 year
  To compared the specificity of combined CTC and ctDNA with those of CTC and ctDNA alone in diagnosis of primary lung cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moon SM, Kim JH, Kim SK, Kim S, Kwon HJ, Bae JS, Lee S, Lee HS, Choi MY, Jeon BH, Jeong BH, Lee K, Kim HK, Kim J, Um SW. Clinical Utility of Combined Circulating Tumor Cell and Circulating Tumor DNA Assays for Diagnosis of Primary Lung Cancer. Anticancer Res. 2020 Jun;40(6):3435-3444. doi: 10.21873/anticanres.14329. PMID 32487642